CLINICAL TRIAL: NCT06254066
Title: An Open-label, Single-arm Study of Adebrelimab Combined With Fluzoparib in HRD-positive HR +/HER2- Advanced Breast Cancer
Brief Title: Adebrelimab Combined With Fluzoparib in HRD-positive HR +/HER2- Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-063
Record Dates: First submitted 2024-02-04; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Female Breast Cancer Patients; Histopathologically Confirmed Advanced HR +/HER2-invasive Breast Cancer; HRD Positive Advanced Breast Cancer
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab+Fluzoparib (Experimental)
  Interventions: Drug: Adebrelimab plus Fluzoparib

INTERVENTIONS:
Drug: Adebrelimab plus Fluzoparib — Adebrelimab combined with Fluzoparib in HRD-positive HR +/HER2- advanced breast cancer

SUMMARY:
This is an open-label, single-arm, exploratory study planned to include 40 patients with HRD-positive HR +/HER2- advanced breast cancer treated with Adebrelimab in combination with fluzoparib. To observe and evaluate the efficacy and safety of Adebrelimab combined with fluzoparib in the treatment of HRD-positive HR +/HER2-advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients aged ≥ 18 years and ≤ 75 years;
2. Histopathologically confirmed advanced HR +/HER2-invasive breast cancer according to the latest ASCO/CAP guidelines, meeting the following conditions: HER2 negative: IHC 0/1 + or IHC2 + but ISH negative; ER positive: IHC ≥ 1%, PR positive: IHC ≥ 1%
3. ECOG score 0 ~ 2;
4. In the treatment stage of recurrence and metastasis, ≤ 1 line of chemotherapy is allowed, at least ≥ 1 standard endocrine therapy (including CDK4/6 inhibitor therapy) is allowed, and ≤ 1 antibody-conjugated drug (ADC) is allowed;
5. HRD positive confirmed, known germline and/or systemic BRCA mutation status and HRR pathway-related gene mutation status allow preferential enrollment;
6. Appropriate level of organ function
7. Patients voluntarily participate in and sign the informed consent form, are expected to have good compliance and cooperate with the study according to the requirements of the protocol.

Exclusion Criteria:

1. Active or symptomatic brain metastases Systemic anticancer therapy (including chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, or tumor embolization) within 14 days prior to enrollment
2. Patients previously received PD-1/PD-L1 antibody, CTLA-4 antibody, or other treatments against PD-1/PD-L1 inhibitors;
3. Female patients who are pregnant and lactating, female patients who are fertile and have a positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial.4.Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia, and the subject has a known history of psychotropic drug abuse, alcoholism

5.Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); positive hepatitis B surface antigen (HBsAg) test, or positive hepatitis B core antibody (HBcAb) test followed by positive HBV-DNA test (HBV-DNA test was performed only in patients with negative HBsAg test and positive HBcAb test); positive hepatitis C virus (HCV) antibody test followed by positive HCV-RNA test (HCV-RNA test was performed only in patients with positive HCV antibody test) 6.Any other condition that, in the opinion of the investigator, would make the patient inappropriate for participation in this study.

Ages: 18 Months to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-16 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 6-10 months
  Progression-free survival

IPD SHARING:
Plan to Share IPD: No